CLINICAL TRIAL: NCT07040800
Title: Adherence to Pharmacotherapy in Patients Admitted for Inpatient Treatment at the Scientific Medical Center
Brief Title: Adherence to Pharmacotherapy in Patients Admitted for Inpatient Treatment at the Scientific Medical Center (PRIMULA)
Status: Active, not recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-06/25
Record Dates: First submitted 2025-06-09; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: drug therapy; medical recommendations; commitment
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional observational study will assess adherence to previously prescribed medication in patients admitted to inpatient treatment at the scientific medical center. When filling out the questionnaire, the previously prescribed pharmacotherapy, the regularity of medication intake and the presence of side effects of drug treatment, if any, according to their medical history will be clarified.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the scientific center, signed patients' informed consent

Exclusion Criteria:

* patient's unsigned informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to a multidisciplinary hospital
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with NSEPh adherence score ≥3 (i.e., complete secondary or complete primary non-commitment) at baseline | Baseline
  Commitment to treatment was determined using the National Society of Evidence-Based Pharmacotherapy (NSEPh) adherence scale.
  Based on the scores obtained, patients are categorized as follows:
  * 0 points - full adherence
  * 1 point - partial (incomplete) non-commitment, unintentional violations
  * 2 points - partial (incomplete) non-commitment, intentional violations (including self-medication)
  * 3 points - complete secondary non-commitment
  * 4 points - complete primary non-commitment The threshold for defining non-adherence was set at ≥3 points.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Centre for Therapy and Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No